CLINICAL TRIAL: NCT01784705
Title: Transcranial Bright Light Therapy in Seasonal Affective Disorder (SAD)- a Randomized Placebo-controlled Trial
Brief Title: Transcranial Bright Light Therapy in Seasonal Affective Disorder (SAD)
Acronym: SAD3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Heidi Jurvelin, Research coordinator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCT-003
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Seasonal Affective Disorder (SAD)
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Transcranial bright light therapy (Experimental)
  Interventions: Device: Transcranial bright light therapy
- Transcranial placebo treatment (Placebo Comparator)
  Interventions: Device: Transcranial placebo treatment

INTERVENTIONS:
Device: Transcranial bright light therapy — The bright light treatment was given transcranially via ear canals by using bright light device. The bright light was produced using two light-emitting diodes (LEDs). The bright light was transmitted into both ear canals by an optical fibre. Daily 12 minutes TBL was taken at home during forenoon.
  Arms: Transcranial bright light therapy
Device: Transcranial placebo treatment — The placebo treatment was given transcranially via ear canals by placebo device. Daily 12 minutes placebo treatment was taken at home during forenoon.
  Arms: Transcranial placebo treatment

SUMMARY:
Bright light therapy (BLT) has been found to be effective in treatment of seasonal affective disorder (SAD). The mechanism of action of conventional BLT in the treatment of SAD is under debate. Recently, transcranial bright light (TBL) via ear canals has been proved to modulate the neural networks of the human brain and improve cognitive performance in healthy subjects. Moreover, TBL has been found to alleviate symptoms of SAD in open trial. In this case the investigators will study the effect of transcranial bright light treatment via ear canals on depressive and anxiety symptoms in patients suffering from SAD in randomized controlled double-blind study design.

ELIGIBILITY:
Inclusion Criteria:

* patient has (according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision [DSM-IV-TR]) a Major depression, recurrent episode, seasonal pattern
* Structured Interview Guide for the Hamilton Depression Rating Scale - Seasonal Affective Disorder Version Self Rating Version (SIGH-SAD-SR) score ≥ 16
* patient is over 18 years and under 66 years
* patient can read and understand the subject information sheet
* patient has signed the informed consent form
* patient is not pregnant

Exclusion Criteria:

* patient has a lifetime psychotic disorder
* patient has a bipolar disorder
* patient has alcohol or some other substance use dependence or misuse
* patient has some unstable somatic disorder
* patient uses some psychotropic agencies
* patient is, in the opinion of the investigator, unsuitable for any reason
* patient is a member of the site personnel or their immediate families
* patient has administered bright light therapy via ear canals during the current episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Structured Interview Guide for the Hamilton Depression Rating Scale - Seasonal Affective Disorder Version Self Rating Version, total score ≤9 | At the end of the four week study period
  Remission, i.e., Structured Interview Guide for the Hamilton Depression Rating Scale - Seasonal Affective Disorder Version Self Rating Version total score ≤ 9

SECONDARY OUTCOMES:
Beck Depression Inventory-II, total score <=10 | At the end of the four week study period
  Remission, i.e.,Beck Depression Inventory-II, total score <=10
State Trait Anxiety Inventory -Y2, total score | At the end of the four week study period
Trail- making test (TMT-A and TMT-B),total time | At the end of the four weeks study period

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University, Oulu, Finland